CLINICAL TRIAL: NCT06002932
Title: Comparison of PROVISIONal 1-stent Strategy with Drug-Eluting Balloon Versus Planned 2-stent Strategy in Patients with Non-LM Coronary True-Bifurcation Lesions.
Brief Title: Comparison of PROVISIONal 1-stent Strategy with DEB Versus Planned 2-stent Strategy in Coronary Bifurcation Lesions.
Acronym: PROVISIONDEB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: XC22EIDI0051
Record Dates: First submitted 2023-07-31; First posted 2023-08-21 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: coronary artery disease; percutaneous coronary intervention; coronary bifurcation lesion; strategy
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional arm (Active Comparator): As per the conventional treatment process, this strategy treats both the main vessel and the branch vessel with stents. The decision among Crush (Mini-crush), DK-Crush, Cullotte, TAP, and T-stenting is left to the discretion of the treatment provider.
  Interventions: Procedure: Procedure: planed 2-stent strategy
- PROVISION-DEB arm (Experimental): As a principal, the treatment regime will be composed of the stent treatment in the main blood vessel and a drug-eluting balloon in a branch vessel. The order of the treatments done to the main vessel and the branch vessel shall be at the discretion of the treatment provider. Also, at the discretion of the treatment provider, a bail-out stenting can still be performed, depending on the condition of the branch vessel following a drug-eluting balloon treatment. However, bail-out stenting is recommended if there is a TIMI flow disorder, severe coronary artery exfoliation (National Heart, Lung, and Blood Institute type D, E, or F), or significant residual stenosis.
  Interventions: Procedure: Procedure: provisional 1-stent plus DEB strategy

INTERVENTIONS:
Procedure: Procedure: planed 2-stent strategy — Procedure: planed 2-stent strategy
  Arms: Conventional arm
Procedure: Procedure: provisional 1-stent plus DEB strategy — Procedure: provisional 1-stent plus DEB strategy
  Arms: PROVISION-DEB arm

SUMMARY:
[The Purpose of the Clinical Study] The purpose of this randomized comparison study is to compare the 1-stent strategy with a drug-eluting balloon and the 2-stent strategy in patients with non-LM coronary true-bifurcation lesions.

[Hypothesis] In this study, the researchers intend to verify the hypothesis that the 1-stent strategy with a drug-eluting balloon is non-inferior to the 2-stent strategy in terms of target lesion failures (cardiac death, target vessel MI, or target vessel revascularization).

DETAILED DESCRIPTION:
1. Provisional 1-stent plus DEB strategy As a principal, the treatment regime will be composed of the stent treatment in the main blood vessel and a drug-eluting balloon in a branch vessel. The order of the treatments done to the main vessel and the branch vessel shall be at the discretion of the treatment provider. Also, at the discretion of the treatment provider, a bail-out stenting can still be performed, depending on the condition of the branch vessel following a drug-eluting balloon treatment. However, bail-out stenting is recommended if there is a TIMI flow disorder, severe coronary artery exfoliation (National Heart, Lung, and Blood Institute type D, E, or F), or significant residual stenosis.
2. Planned 2-stent strategy As per the conventional treatment process, this strategy treats both the main vessel and the branch vessel with stents. The decision among Crush (Mini-crush), DK-Crush, Cullotte, TAP, and T-stenting is left to the discretion of the treatment provider.

ELIGIBILITY:
Inclusion Criteria:

① 19+ years old

② Patients with the following lesions and clinical factors. 2-1. The lesion factor: Visually confirmed diameter of the 2.25-2.75 mm in branched vessels, where the main blood vessel's diameter is at least 2.5 mm; the lesion at the branched vessels is of a Medina classification (1,1,1), (1,0,1), or (0,1,1), with a true bifurcation; a de novo lesion.

2-2 Clinical factors: Stable angina pectoris, unstable angina pectoris, or myocardial infarction with an elevated non-ST segment, all at least 24 hours after their last treatment.

③ Patients who understood the definitions of the test group and the control group and the risks involved in the treatment, and with voluntary, informed consent to participate in the study, as provided either by the patient or their legal representatives.

Exclusion Criteria:

* Patients with myocardial infarction involving an elevated ST segment, or patients with an LM coronary true-bifurcation lesion.

  * Patients who are ruled out by the treatment provider because the 2-stent strategy was deemed unsuitable to the patient due to a clinical condition.

    * A patient with aspirin or P2Y12 inhibitors (ticagrelor or clopidogrel) contraindications.

      * A patient who experienced psychogenic shock at the time of admission, or showed severe left ventricle insufficiency (where the left ventricle ejection fraction is less than 30%.)

        * A patient who requires prolonged anti-coagulative treatment (warfarin or a new oral anti-coagulant [NOAC])

          * A patient who is currently hemorrhagic, or has a high risk of major hemorrhage (active peptic ulcer, GI lesions with high hemorrhagic risks, malicious tumors with a high risk of hemorrhage) ⑦ A patient with a history of intra-cerebral hemorrhage or intra-cerebral aneurysm.

            * A patient for whom surgery that requires antiplatelet treatment intervention is scheduled within the next six months.

              ⑨ A patient with severe hepatic diseases (abdominal effusion) Platelet count at less than 80,000 cells/mm3 Hgb count at less than 10 g/dL

              ⑩ A patient who appears to be at risk of bradycardia (a patient with an insufficiency of the said function, or a patient without a permanent pacemaker despite a grade 2 or higher atrioventricular block).

              ⑪ A patient who tested positive in a pregnancy test, or is currently breastfeeding

              ⑫ A patient with less than one year of remaining life expectancy due to comorbidity (based on the medical judgment of the investigator).

              ⑬ A patient who is already participating in another randomized clinical study for other medicines or medical devices, where the primary end point has not been reached.

              ⑭ A patient who did not sign her informed consent form, or could not be traced in the long-term.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
target lesion failure the number of events | 12 months after randomization
  composite outcomes the number of events (cardiac death, target vessel myocardial infarction, or ischemia-driven target lesion revascularization)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Ho Her, MD. PhD., Principal Investigator — St Vincent's Hospital
Locations (1):
- St. Vincent's Hospital , the Catholic University, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No